CLINICAL TRIAL: NCT05432336
Title: Complex Ocular Infection, Optimization of Microbiological Diagnosis
Acronym: ICODIA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220259; 2021-A02587-34 (Other: France : ANSM)
Record Dates: First submitted 2022-05-12; First posted 2022-06-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Endophthalmitis; Keratitis
Keywords: Endogenous Endophtalmitis; exogenous endophtalmitis; keratitis; PCR; NGS
MeSH Terms: conditions — Endophthalmitis; Keratitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Complex ocular infections (COI): All patients with an COI (endophtalmitis or hospitalized keratitis)
  Interventions: Diagnostic Test: NGS for endohtalmitis / Multiplex PCR for keratitis

INTERVENTIONS:
Diagnostic Test: NGS for endohtalmitis / Multiplex PCR for keratitis — For endophtalmitis : optimizing culture and NGS will be realized
  For keratitis: Multiplex PCR will be added on ocular samples
  Other Names: Bundle of intervervention to optimizing diagnosis of ocular complex infections

SUMMARY:
The purpose of this study is to evaluate the impact of different technique to optimize the microbiological diagnosis of the COI.

* Metagenomic for the endophtalmitis
* Multiplex polymerase chain reaction for corneal abscesses

DETAILED DESCRIPTION:
Microbiological diagnosis of complex ocular infection (COI) (i.e: endophtalmitis and corneal abscess) is a current challenge. Indeed, endophtalmitis are often germ-free because a lack of microbiological diagnosis due to small volume to analyze and a complex site to attain. The microbiological etiologies of corneal abscesses are more frequently identified.

Since few years, new molecular tools are developed in infectious diseases to optimizing the microbiological diagnosis. The investigators implemented these techniques in our hospital to optimize the microbiological diagnosis of complex ocular infection (COI). Thus, endophtalmitis benefit, when the volume of the ocular sample is sufficient, of molecular techniques (16s PCR and metagenomic shotgun). Corneal abscesses could shortly benefit of multiplex PCR in order to reduce the time to diagnosis.

The impact and accuracy of these techniques is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient presenting or having presented a clinical suspicion of complex ocular infection requiring a sample for microbiological diagnosis:

  * Corneal abscess requiring hospitalization
  * Any suspicion of endogenous or exogenous endophthalmitis.
* Patient not opposed to participating in the research

Exclusion Criteria:

* Patient under guardianship or curatorship
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient presenting or having presented a clinical suspicion of complex ocular infection requiring a sample for microbiological diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Positivity rates of COI samples according to the new protocol | 2 weeks after taking samples
  Before/after type comparison. Comparison of the positivity rates of COI samples according to the new protocol: (i) for endophthalmitis performing a vitreous puncture (PV) or an anterior chamber puncture (PCA), or corneal scraping, optimized with modification of microbiological techniques (culture on enriched medium alone associated with shotgun metagenomics), (ii) for severe corneal abscesses, addition to standard microbiological techniques of molecular biology tests (multiplex PCR and / or metagenomics).
  An COI will be considered with a positive microbiological diagnosis after multidisciplinary concertation considering the different results

SECONDARY OUTCOMES:
Microbiological diagnosis of the infection | At the end of the follow up: 18 months
  Analysis of a prospective cohort of COI
Time to microbiological diagnosis according to the different technic | At the end of the follow up: 18 months
  Analysis of a prospective cohort of COI
Accuracy of the different technics according to the gold standard (microbiological culture) | At the end of the follow up: 18 months
  Analysis of a prospective cohort of COI
Visual acuity | At the end of the follow up: 18 months
  Evaluation of visual acuity at the end of treatment and the cure rate. The investigators hypothesized that the improvement of the microbiological diagnosis allows an improvement of the therapeutic management and thus of the visual outcome.
Cure rate | At the end of the follow up: 18 months
  Evaluation of visual acuity at the end of treatment and the cure rate. The investigators hypothesized that the improvement of the microbiological diagnosis allows an improvement of the therapeutic management and thus of the visual outcome.
Modification or not of the anti-infectious treatment | At the end of the follow up: 18 months
  Analysis of the impact of microbiological diagnosis on the choice of anti-infectious molecules..
  The investigators hypothesized that the improvement of the microbiological diagnosis and the implementation of the COI management bundle will induce a modification of the prescription of anti-infectious molecules. The investigators will realize a qualitative and quantitative analysis of prescribed anti-infective molecules

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CANOUI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Equipe mobile d'infectiologie, Cochin hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided